CLINICAL TRIAL: NCT03249558
Title: Effect of Combined Morphine and Duloxetine on Chronic Pain
Acronym: Duloxetine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Vice Chair for Research; Chief, Division of Pain Medicine; Director, MGH Center for Translational Pain Research, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2017P001589
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Chronic Low Back Pain; Chronic Neck Pain
Keywords: Pain; Pain Management
MeSH Terms: conditions — Pain; Agnosia | interventions — Morphine; Duloxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Morphine, Duloxetine (Active Comparator): Subjects will take a maximum dose of 60 mg/day of extended release morphine capsules and 60 mg of duloxetine capsules.
  Interventions: Drug: Morphine; Drug: Duloxetine
- Morphine, Placebo Duloxetine (Placebo Comparator): Subjects will take a maximum dose of 60 mg/day of extended release morphine capsules and placebo duloxetine capsules.
  Interventions: Drug: Morphine; Drug: Placebo
- Placebo Morphine, Duloxetine (Placebo Comparator): Subjects will take placebo morphine capsules and 60 mg of duloxetine capsules.
  Interventions: Drug: Duloxetine; Drug: Placebo

INTERVENTIONS:
Drug: Morphine — Subjects will be randomized into one of the treatment groups and will follow the assigned medication schedule for 10 weeks. Quantitative Sensory Testing (QST) will be performed on the subjects to compare pain threshold, pain tolerance, and wind up.
  Other Names: Morphine Sulfate Contin, Morphine Sulfate Instant Release
  Arms: Morphine, Duloxetine; Morphine, Placebo Duloxetine
Drug: Duloxetine — Subjects will be randomized into one of the treatment groups and will follow the assigned medication schedule for 10 weeks. Quantitative Sensory Testing (QST) will be performed on the subjects to compare pain threshold, pain tolerance, and wind up.
  Other Names: Cymbalta
  Arms: Morphine, Duloxetine; Placebo Morphine, Duloxetine
Drug: Placebo — Subjects will be randomized into one of the treatment groups and will follow the assigned medication schedule for 10 weeks. Quantitative Sensory Testing (QST) will be performed on the subjects to compare pain threshold, pain tolerance, and wind up.
  Other Names: Sugar pill
  Arms: Morphine, Placebo Duloxetine; Placebo Morphine, Duloxetine

SUMMARY:
A double-blind, randomized, and placebo-controlled clinical study examining whether duloxetine, a serotonin and norepinephrine reuptake inhibitor (SNRI), could enhance opioid analgesia and reduce overall opioid use. Positive outcomes will help improve the overall effectiveness of clinical opioid therapy and reduce unnecessary opioid dose escalation.

DETAILED DESCRIPTION:
Subjects will participate in a 10-week study consisting of three phases: Phase I is the dose titration period of 4 weeks, Phase II is the dose maintenance period of 4 weeks, and Phase III is the dose taper period of 2 weeks. Seven office visits (Initial visit/baseline, weeks 1, 3, 5, 7, 9, and end of week 10) and four follow up phone calls (weeks 2, 4, 6, and 10) will be used to collect data. Since this is a prospective study, we will be able to first determine baseline QST and VAS pain score, followed by assessing their longitudinal changes at each office visit. To assess OIH, QST will be performed at each office visit before subject takes the next dose of the study drugs. We will also measure plasma morphine concentration during the titration and maintenance phase to help validate morphine intake.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18-70 years old.
2. Subject has chronic neck or back pain for at least 3 months.
3. Subject has a VAS ≥ 5.
4. Has not taken duloxetine in the last 3 months.
5. Has not taken an opioid in the last 3 months, but has taken one in the past without sufficient pain control OR has never taken opioids but has failed at 3 (or more) non-opioid treatments.

Exclusion Criteria:

1. Subject has major psychiatric disorders requiring recent hospitalization (within 3 months) such as major depression, bipolar disorder, schizophrenia, anxiety disorder, or psychotic disorder.
2. Subject is using illicit drugs detected by urine toxicology/drug screen.
3. Subject is pregnant or lactating/breast feeding.
4. Subject is allergic to morphine or duloxetine.
5. Subject is on an antidepressant including serotonin-norepinephrine reuptake inhibitors (SNRI), selective serotonin reuptake inhibitor (SSRI), tricyclic antidepressant.
6. Subject has a history of suicidal attempts or current suicidal ideation.
7. Subject takes monoamine oxidase inhibitors, antipsychotics, triptan drugs such as sumatriptan, lithium, linezolid, tramadol (Ultram), St. John's Wort, central nervous system (CNS) stimulants such as amphetamine, methylphenidate, methamphetamine, phentermine, diethylpropion, sibutramine, cocaine, or thioridazine.
8. Subject has uncontrolled narrow-angle glaucoma.
9. Subject has sensory deficits on arms or Raynaud's Syndrome.
10. Subject has a pending litigation related to chronic pain condition.
11. Subject is on methadone or suboxone treatment for addiction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Karina de Sousa, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Massachusetts General Hospital Center for Translational Pain Research — https://www.massgeneral.org/anesthesia/translational-pain-research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment goal was not met by the planned completion time.
Pre-assignment Details: 81 participants were consented to this study. 22 were not randomized to one of 3 groups as they were deemed ineligible to continue or withdrew from the study. 59 were randomized to 1 of 3 groups. 28 of which completed the study.
Period: Overall Study
Arm/Group | Morphine, Duloxetine | Morphine, Placebo Duloxetine | Placebo Morphine, Duloxetine
Started | 21 | 19 | 19
Completed | 10 | 12 | 6
Not Completed | 11 | 7 | 13
Not completed — Lost to Follow-up | 2 | 1 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 7
Not completed — COVID-19 pandemic shutdown | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: 81 participants were consented. 22 were deemed ineligible to continue after screening so only 59 were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine, Duloxetine | Morphine, Placebo Duloxetine | Placebo Morphine, Duloxetine | Total
Number analyzed (Participants) | 21 | 19 | 19 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 17 | 46
  >=65 years | 8 | 3 | 2 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 19
  Male | 14 | 13 | 13 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 1 | 7
  Not Hispanic or Latino | 19 | 15 | 17 | 51
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 7 | 18
  White | 13 | 10 | 8 | 31
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Opioid Dose (Morphine-equivalent Dose in mg)
Description: The investigators will compare overall opioid dose (in morphine-equivalent dose in mg) between the morphine/duloxetine group and the morphine/placebo group and compare rescue dose among all three groups. The higher overall opioid dose, the more consumption of opioid.
Time Frame: 10 weeks
Population: The data collection was incomplete for the subjects who completed the study, therefore, the summary can not be provided. The total number of participants needed for analysis was not reached, and the results information provided are regarding the subjects who completed the study.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Morphine, Duloxetine | Morphine, Placebo Duloxetine | Placebo Morphine, Duloxetine
Number analyzed (Participants) | 21 | 19 | 19
mg | 19.6 (2.05) | 19.6 (2.16) | 19.6 (2.16)

2. Primary Outcome: Visual Analog Scale (VAS)
Description: To examine changes in pain intensity measured on a Visual Analog Scale with units on a scale ranging from 0 cm-10 cm (0 cm being lowest and 10 cm being the higher the score, where values closer to 10 cm reflect more pain) and to determine total versus rescue opioid use after each treatment.
Time Frame: 10 weeks
Population: The data collection was incomplete for the subjects who completed the study, therefore, the summary and outcome can not be provided. The total number of participants needed for analysis was not reached, and the results information provided are regarding the subjects who completed the study. Due to the total number of participants needed for analysis not being met, the summary can not be provided.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Morphine, Duloxetine | Morphine, Placebo Duloxetine | Placebo Morphine, Duloxetine
Number analyzed (Participants) | 10 | 12 | 6
cm | 2.8 (3.05) | 2.33 (3.05) | 4.66 (3.05)

ADVERSE EVENTS:
Time Frame: The adverse events were monitored and assessed through study completion, an average of 6 months.
Description: Definition does not defer.
Arm/Group | Morphine, Duloxetine | Morphine, Placebo Duloxetine | Placebo Morphine, Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
In this study we did not enroll enough participants to reach the number needed for our analysis to have power which is a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03249558/Prot_SAP_000.pdf